CLINICAL TRIAL: NCT01925664
Title: Doula Support for Young Mothers: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R40 MC 00203
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Parenting; Breastfeeding; Depression, Postpartum
Keywords: Doulas; Parenting; Breastfeeding; Pregnancy in Adolescence
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum | interventions — Doulas

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doula (Experimental): Mothers received doula home visiting services in addition to normal prenatal and obstetric clinical care and had access to social work case management.
  Interventions: Behavioral: Doula
- Usual Care (No Intervention): Mothers received normal prenatal and obstetric clinical care and had access to social work case management.

INTERVENTIONS:
Behavioral: Doula — This intervention included doulas providing weekly home visits during the last trimester of pregnancy and up to three months postpartum. Home visits focused on prenatal health, preparation for childbirth, breastfeeding education, and developing a relationship with the baby. Doulas also were present in the hospital during labor, delivery, and postpartum providing emotional support, non-medical comfort measures, and breastfeeding counseling.
  Arms: Doula

SUMMARY:
The goal of this study was to evaluate the impact of a doula home visiting intervention on young, low-income mothers' birth outcomes, breastfeeding, postpartum depressive symptoms, and parenting, and on their children's development.

DETAILED DESCRIPTION:
The goal of this study is to evaluate a doula home visiting model -- sometimes called the "community doula model." This model differs from typical hospital based doula interventions in several ways. Doulas are providers from the same community backgrounds as their clients. Services are not just provided during labor and delivery, but throughout the final trimester and during the first weeks after delivery. Prenatal and postpartum services are provided in the homes of the mothers. The model was developed specifically for working with low-income mothers and with young mothers.

A two-armed randomized controlled trial was conducted at the University of Chicago Hospitals. Participants were recruited through two out-patient obstetric clinics affiliated with the Hospitals. The clinics primarily served a low-income, African-American population, reflective of the families in the communities near to the hospital. The study was open to all young women receiving prenatal care at the clinics who met age and eligibility criteria. After providing informed consent and completing a baseline interview, participants were randomized into two groups. The experimental group, in addition to receiving regular clinical care, received weekly home visiting services from a doula and the support of a doula at the hospital during labor and delivery. Doulas worked with their clients until three months postpartum. The control group received standard clinical care and had access to social work case management.

Four paraprofessional doulas delivered the study intervention. Before providing study services, doulas had been trained to provide childbirth education, labor support, breastfeeding education, and parent-child interaction support.

Followup research assessments of the doula and control group mothers and infants were conducted during the first three days postpartum, at 4 months postpartum, at 12 months postpartum, and at 24 months postpartum. 80% of the sample was retained through the 24 month followup assessment. Follow up assessments involved interviews with the mothers, videotaping of mother-infant interaction, and behavioral assessment of the infants. Obstetric and newborn hospital medical charts were also reviewed.

The study evaluated outcomes that have been the focus of prior studies of hospital-only doula services: use of obstetrical intervention in labor and delivery (anesthesia, surgical delivery), mother labor efficacy, breastfeeding, and maternal depression. A major contribution of this study is to explore longer term outcomes not evaluated in prior studies of doula intervention, particularly parenting and child development outcomes. The study evaluated multiple dimensions of parenting including parenting behavior (sensitivity, stimulation), parenting efficacy, parenting attitudes, and parenting stress. Child development outcomes included cognitive development and early behavior problems.

ELIGIBILITY:
Inclusion Criteria:

* pregnant and less than 34 weeks gestation
* planning to deliver at study hospital
* between ages 14 and 21

Exclusion Criteria:

* planning to move out of community after giving birth
* planning to give up custody of infant
* prior c-section delivery

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 248 (Actual)
Dates: Start 2001-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Initiation | Three days postpartum
Positive parenting behavior (Parent Child Observation Guide) | 4 months postpartum
  Videotaped interactions between mothers and infants coded by masked observers

SECONDARY OUTCOMES:
Breastfeeding duration | 4- and 12 months postpartum
Positive parenting behaviors (Parent Child Observation Guide) | 12- and 24 months postpartum
  Videotaped interactions between mothers and infants coded by masked observers
Use of labor anesthesia | Start of labor through childbirth
Labour Agentry Scale | 1 day postpartum
  The Labour Agentry Scale is a self-report scale that assesses maternal feelings of efficacy during labor
Adult Adolescent Parenting Inventory (AAPI) | 4 months postpartum
  The AAPI is a self report scale that measures appropriate parenting attitudes
Maternal Self-Efficacy Scale | 4-, 12-, and 24 months postpartum
  The Maternal Self-Efficacy Scale is a self report scale that measures parenting efficacy with regard to infant care.
Parenting Stress Index (PSI) | 4-, 12-, and 24 months postpartum
  The PSI is a self report scale that measures parenting stress and parent perceptions of the difficulty of her child
Center for Epidemiologic Studies Depression Scale (CES-D) | 4-, 12-, and 24 months postpartum
  The CES-D is a self report scale that measures depressive symptoms experienced in the prior week.
Timing of solid food introduction to infant | 4- and 12 months postpartum
The Brief Infant Toddler Social Emotional Assessment (BITSEA) | 12- and 24 months postpartum
  The BITSEA is a parent report measure that assesses problem behaviors and social competence in infants and toddlers.
Mullen Scales of Early Learning | 24 months postpartum
  The Mullen is an assessment tool that measures child motor, cognitive, and language development. Trained assessors administered the instrument to the toddlers of study mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Sydney L Hans, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Edwards RC, Thullen MJ, Korfmacher J, Lantos JD, Henson LG, Hans SL. Breastfeeding and complementary food: randomized trial of community doula home visiting. Pediatrics. 2013 Nov;132 Suppl 2:S160-6. doi: 10.1542/peds.2013-1021P. PMID 24187119